CLINICAL TRIAL: NCT05882175
Title: A Prospective Study to Validate the Prognostic Power of the Optimized HLH Inflammatory (OHI) Index
Brief Title: Prospective Validation of the OHI Index
Acronym: HLH
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Rabin Medical Center (Other); Sheba Medical Center (Other Government); Schneider Children's Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 0321-19-MMC
Record Dates: First submitted 2021-01-19; First posted 2023-05-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: HLH; Hemophagocytic Lymphohistiocytoses; Hemophagocytic Syndrome; Hematologic Malignancy; Hematologic Neoplasms
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples and peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OHI+ patients: Adult patients with hematologic malignancies that have sCD25>3,900 U/mL and ferritin >1,000 ng/mL
- OHI- patients: Adult patients with hematologic malignancies, with sCD25>3,900 U/mL and/or ferritin < 1,000 ng/mL

SUMMARY:
Hemophagocytic lymphohistiocytosis (HLH) associated with hematologic malignancies (HM-HLH) is a syndrome with an abysmal prognosis (10-30% 5 years overall survival). The investigators have recently established an improved diagnostic and prognostic index for HM-HLH, termed the Optimized HLH Inflammatory (OHI) index. The OHI index is comprised of the combined elevation of soluble CD25 (sCD25) > 3,900 U/mL and ferritin >1,000 ng/mL . However, the true incidence and outcomes of HLH/OHI+ in an unselected cohort are unknown, and so is the mechanism of HM-HLH.

DETAILED DESCRIPTION:
The investigators will enroll patients with new/transformed hematologic malignancies. The investigators will follow the patients until the end of the study, report their survival at one year and examine their prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies
* At least 18 years old

Exclusion Criteria:

* Prior recent treatment (chemotherapy/ other cytoreductive therapies in the last month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and females with new diagnosis/transformation/reactivation of hematologic malignancies
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2030-03-03 (Estimated); Study Completion 2030-03-03 (Estimated)

PRIMARY OUTCOMES:
To assess 365 days mortality of OHI+ and OHI- patients | Mortality rate one year from OHI assessment
  The investigators will use Kaplan-Meier curves to compare survival between OHI+ and OHI- patients

SECONDARY OUTCOMES:
To determine the incidence of OHI+ patients in our cohort | The investigators will assess the incidence after three years of enrollment
  The investigators will assess the incidence of OHI+ within our cohort (OHI+/total patients enrolled)

CONTACTS AND LOCATIONS:
Overall Officials: Adi Zoref-Lorenz, Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zoref-Lorenz A, Murakami J, Hofstetter L, Iyer S, Alotaibi AS, Mohamed SF, Miller PG, Guber E, Weinstein S, Yacobovich J, Nikiforow S, Ebert BL, Lane A, Pasvolsky O, Raanani P, Nagler A, Berliner N, Daver N, Ellis M, Jordan MB. An improved index for diagnosis and mortality prediction in malignancy-associated hemophagocytic lymphohistiocytosis. Blood. 2022 Feb 17;139(7):1098-1110. doi: 10.1182/blood.2021012764. PMID 34780598